CLINICAL TRIAL: NCT05778058
Title: he Effect of Transcutaneous Auricular Vagus Nerve Stimulation on Cycling Ergometry and Recovery in Healthy Young Individuals
Brief Title: The Effect of Vagus Nerve Stimulation on Cycling Ergometry and Recovery
Acronym: TAVNSCER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sinop University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: VNS003
Record Dates: First submitted 2021-09-15; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Healthy; Sports Physical Therapy; Activity, Motor
Keywords: Vagus Nerve Stimulation; Physiological Parameters; Recovery; Cycle Ergometer Test; Transcutaneous Auricular
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: 90 healthy young individuals were included in the study. Participants were randomly divided into 3 groups as unilateral (n=30, 15 female, 15 male), bilateral (n=30, 15 female, 15 male) and bilateral sham (n=30, 15 female, 15 male) groups. ). The cycling exercise was performed at maximum performance for 30 minutes under the same wattage load. Non-invasive ear stimulation was performed with the Vagustim device according to the participant groups. Pulse, systolic and diastolic blood pressure, distance, pain, fatigue, lactic acid level and autonomic nervous system were evaluated before, after and at the end of cycling exercise. Oneway Anova test and Kruskal Wallis test were used between groups. Dunn's test was used to determine the group that caused the difference. Analysis of variance was used for repeated measurements, Bonferroni test and Friedman test were used for in-group comparisons. Significance was evaluated at the p<0.05 level.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Unilateral Stimulation (Experimental): After evaluating with 7 different parameters on the first, second, third and fourth days of the protocol, the participants in all groups will be asked to do cycling exercise with maximum performance for 30 minutes under the same wattage load.
  It will be re-evaluated after the cycling exercise application. After the assessment is complete, stimulation will be given with Vagustim non-invasively for 30 minutes. After vagus nerve stimulation, a re-evaluation will be made and the protocol for that day will be terminated.
  With the Vagustim device, vagus nerve stimulation will be applied in one ear for 20 minutes, with a frequency of 10 Hz, a pulse width of 300 μs in Modulation mode, and a constant current that the participant will feel the current comfortably.
  Interventions: Device: Unilateral Stimulation; Diagnostic Test: Bicycle Ergometer Test; Diagnostic Test: Lactat Scout; Diagnostic Test: Polar H10; Device: Vagustim Device
- Bilateral Stimulation (Experimental): After evaluating with 7 different parameters on the first, second, third and fourth days of the protocol, the participants in all groups will be asked to do cycling exercise with maximum performance for 30 minutes under the same wattage load.
  It will be re-evaluated after the cycling exercise application. After the assessment is complete, stimulation will be given with Vagustim non-invasively for 20minutes. After vagus nerve stimulation, a re-evaluation will be made and the protocol for that day will be terminated.
  With the Vagustim device, vagus nerve stimulation will be applied in bilateral ear for 20 minutes, with a frequency of 10 Hz, a pulse width of 300 μs in Modulation mode, and a constant current that the participant will feel the current comfortably.
  Interventions: Device: Bilateral Stimulation; Diagnostic Test: Bicycle Ergometer Test; Diagnostic Test: Lactat Scout; Diagnostic Test: Polar H10; Device: Vagustim Device
- Bilateral Sham Stimulation (Sham Comparator): After evaluating with 7 different parameters on the first, second, third and fourth days of the protocol, the participants in all groups will be asked to do cycling exercise with maximum performance for 30 minutes under the same wattage load. Bisiklet egzersiz uygulaması sonrasında tekrar değerlendirilecektir.
  It will be re-evaluated after the cycling exercise. After the assessment is complete, sham stimulation with Vagustim for 20 minutes will be given non-invasively. After vagus nerve stimulation, a re-evaluation will be made and the protocol for that day will be terminated.
  Interventions: Device: Bilateral Sham Stimulation; Diagnostic Test: Bicycle Ergometer Test; Diagnostic Test: Lactat Scout; Diagnostic Test: Polar H10; Device: Vagustim Device

INTERVENTIONS:
Device: Unilateral Stimulation — With the Vagustim device, vagus nerve stimulation will be applied in one ear for 20 minutes, with a frequency of 10 Hz, a pulse width of 300 μs in Modulation mode, and a constant current that the participant will feel the current comfortably.
  Arms: Unilateral Stimulation
Device: Bilateral Stimulation — With the Vagustim device, vagus nerve stimulation will be applied in one ear for 20 minutes, with a frequency of 10 Hz, a pulse width of 300 μs in Modulation mode, and a constant current that the participant will feel the current comfortably.
  Arms: Bilateral Stimulation
Device: Bilateral Sham Stimulation — Participants were shown that the device was working, but no current was given.
  Arms: Bilateral Sham Stimulation
Diagnostic Test: Bicycle Ergometer Test — Participants in this group were asked to perform bicycle exercise with maximum performance under 30 watts for 30 minutes.
Diagnostic Test: Lactat Scout — For lactic acid analysis measurement, the middle fingertip of the athlete is disinfected with an alcohol swab and a blood sample is taken by puncturing the finger.The measuring range is 0.5 - 0.25 mmol/L.
Diagnostic Test: Polar H10 — RR times transferred to computer with Polar H10 are used in heart rate variability analysis. Heart rate data will be transferred to the Kubios program and heart rate variability parameters will be calculated and data on the autonomic nervous system (RMSSD, PNS index, Stress index, SNS index, pNN50, Power LF, Power HF and LF/HF ratio) will be obtained.
Device: Vagustim Device — Vagustim Health Technologies Vagus stimulator device is used for this experiment.

SUMMARY:
It is aIt is aimed to examine the possible benefits and effects of the use of Transcutaneous Auricular Vagus Nerve Stimulation to be applied in healthy individuals for sportive purposes on recovery and sportive performance level.

DETAILED DESCRIPTION:
The 90 people between the ages of 18-35 will be included in the study. Each participant will be randomly divided into 3 groups to be homogeneous after the necessary calculations are made by evaluating with age, gender, weight, height and body mass index before starting the study.

The groups are; It will be in the form of Unilateral Stimulation (n=30), Bilateral Stimulation (n=30) and Bilateral Sham Stimulation (n=30) groups.

After the initial assessment, participants in all groups will be asked to do 30 minutes of cycling exercise at maximum performance under the same wattage load. Cycling will be re-evaluated after exercise. After the assessment is complete, stimulation will be given with Vagustim for 20 minutes non-invasively. After vagus nerve stimulation, a re-evaluation will be made and the protocol for that day will be terminated.

After the pain and fatigue rating scale, the evaluation will be completed by determining the lactate level in the blood with the Lactat Scout. Vagus nerve stimulation will be applied with the Vagustim device for 20 minutes, keeping it biphasic, with a frequency of 10 Hz, a pulse width of 300 μs in Modulation mode, and a constant current where the participant feels the current comfortably.

At the end of the Cycling Ergometer Test and Vagus nerve stimulation, the Autonomic Nervous System, pulse and blood pressure will be evaluated with Polar H10 within 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals between the ages of 18-35,
* Willingness to participate in the study
* Having signed the informed consent form

Exclusion Criteria:

* Cases do not want to continue the study.
* Having regular sports habits or starting in the working process,
* Having a disease related to the respiratory system and starting to use drugs
* Having a disease related to the cardiac system and starting to use drugs
* Presence of any chronic disease and using a drug related to it

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of autonomous parameters | In the 4-day protocol, it was measured 12 times in total, before and after vagus therapy with the bicycle ergometer test.
  Systolic / diastolic blood pressure (mmHg) will be measured with the Braun sphygmomanometer.
Numerical Fatigue Rating Scale | In the 4-day protocol, it was measured 12 times in total, before and after vagus therapy with the bicycle ergometer test.
  The fatigue NRS is a patient-administered, single-item, 11-point horizontal scale anchored at 0 and 10, with 0 representing 'no fatigue' and 10 representing 'as bad as you can imagine'. Patients are asked to 'please rate your fatigue (weariness, tiredness) by selecting the number.
Numerical Pain Rating Scale | In the 4-day protocol, it was measured 12 times in total, before and after vagus therapy with the bicycle ergometer test.
  Pain intensity is frequently measured on an 11-point pain intensity numerical rating scale (PI-NRS), where 0=no pain and 10=worst possible pain.
Bicycle Ergometer Test | It was measured 4 times in aggregation in the 4-day protocol.
  All participants will be asked to perform cycling exercise at maximum performance for 30 minutes under a load of 30 watts. Then, the distance (meters) covered during the exercise will be evaluated for the sportive performance of the participants.
Lactat Scout | It was measured 4 times in total on the 1st and 2nd days of the 4-day protocol.
  For lactic acid analysis measurement, the middle fingertip of the athlete is disinfected with an alcohol swab and a blood sample is taken by puncturing the finger.The measuring range is 0.5 - 0.25 mmol/L.
Polar H10 | It was measured 4 times in total on the 1st and 2nd days of the 4-day protocol.
  RR times transferred to computer with Polar H10 are used in heart rate variability analysis. Heart rate data will be transferred to the Kubios program and heart rate variability parameters will be calculated and data on the autonomic nervous system (RMSSD, PNS index, Stress index, SNS index, pNN50, Power LF, Power HF and LF/HF ratio) will be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: SEFA HAKTAN HATIK, Asst. Prof, Study Director — Sinop University
Locations (1):
- Sefa Haktan Hatik, Sinop, Turkey (Türkiye)